CLINICAL TRIAL: NCT03089931
Title: Change of Lumbar Symptom After Surgical Treatment for Patients With Cervical Stenosis
Acronym: LBP
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chi Heon Kim, Professor, Seoul National University Hospital
Other Study IDs: CSMLBP
Record Dates: First submitted 2017-03-15; First posted 2017-03-24 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Cervical Myelopathy Spondylosis; Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cervical spinal surgery — Cervical laminoplasty or anterior discectomy and fusion

SUMMARY:
Low back pain may be reduced after cervical spinal surgery

DETAILED DESCRIPTION:
The improved back pain score after cervical spinal surgery would be higher than that after non-surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* all patients with cervical myelopathy and low back pain

Exclusion Criteria:

* previous surgery at the lumbar spine
* malignancy
* previous surgery at the cervical spine

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with cervical myelopathy and low back pain
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-11-11 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Low back pain | postoperative 6 months
  improve visual analogue pain score (VAS) more than 1.2/10
functional outcome | postoperative 6 months
  improve Oswestry diability index (ODI) more than 6.2/45

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: No